CLINICAL TRIAL: NCT03014661
Title: Untersuchung Zur Erfassung Und Kontrolle Der Lebensqualität Unter Einer Therapie Mit Pollinex Quattro Bei Heuschnupfen
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Claudia Pföhler, Prof. Dr., Universität des Saarlandes
Other Study IDs: PQ-HOM-001
Record Dates: First submitted 2017-01-02; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: pollinosis, quality of life, specific immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Pollinex Quattro

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group study: Single Group study investigating retrospectively the Quality of life of patients with pollinosis under or after specific immunotherapy with Pollinex quattro
  Interventions: Other: Quality of life under or after therapy with Pollinex quattro

INTERVENTIONS:
Other: Quality of life under or after therapy with Pollinex quattro — To measure Quality of life using the DLQI-index in year one, year two, year three or six month after therapy with Pollinex quattro plus.

SUMMARY:
Questionnaire to measure and control the quality of life of patients with hay fever who are treated or were treated with Pollinex quattro

DETAILED DESCRIPTION:
Questionnaire including 19 questions concerning the Quality of life of patients with hayfeyer under or after therapy with a specific immuntherapy with Pollinex quattro

ELIGIBILITY:
Inclusion Criteria:

* Pollinosis/seasonal Rhinitis based on an allergy against birch/alder/Hazel pollen OR grass/rye pollen OR mugwort
* Therapy with Polinex quattro

Exclusion Criteria:

* Age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult persons with hayfever treated with a specific immunotherapy with Pollinex quattro plus (Allergens: birch/alder/Hazel or grass/rye or mugwort)
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire (DLQI) | during year one, year two, year three of therapy or within 6 months after completion of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Saarland University Hospital. Department of Dermatology, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No